CLINICAL TRIAL: NCT01968850
Title: Bone Antiresorptive Therapy With Antiretroviral Initiation (BATARI) Pilot Trial
Acronym: BATARI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: CIHR Canadian HIV Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CTNPT 021
Record Dates: First submitted 2013-10-09; First posted 2013-10-24 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: HIV
Keywords: osteoporosis; HIV; bone Mineral Density; alendronate; vitamin D
MeSH Terms: conditions — Osteoporosis | interventions — Alendronate; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- no bone anti-resorptive therapy (No Intervention): (standard of care)
- 24-week tx of alendronate/vitamin D (Experimental): Concomitant initiation of a 24 week course of co-formulated alendronate/vitamin D
  Interventions: Drug: alendronate/vitamin D
- Delayed 24-week tx of alendronate/vitamin D (Experimental): a 24 week delay in initiation of a 24 week course of alendronate/vitamin D
  Interventions: Drug: alendronate/vitamin D

INTERVENTIONS:
Drug: alendronate/vitamin D — once weekly 70mg oral dose of alendronate co-formulated with 5600IU vitamin D3 (cholecalciferol) for 24 weeks.
  Other Names: Fosavance 70/56
  Arms: 24-week tx of alendronate/vitamin D; Delayed 24-week tx of alendronate/vitamin D

SUMMARY:
This is a two-site, three-arm, open-label, pilot randomized controlled trial of bone anti-resorptive therapy during ART initiation in HIV-infected adults. Thirty (30) treatment-naïve HIV-infected adults initiating eligible first-line ART regimens will be randomized in a 1:1:1 fashion to one of the following three arms:

1. no bone anti-resorptive therapy (standard of care)
2. concomitant initiation of a 24 week course of co-formulated alendronate/vitamin D;
3. a 24 week delay in initiation of a 24 week course of alendronate/vitamin D

Assessments (including clinical evaluation, questionnaires, adherence, basic laboratory evaluation, and BMD measurement) will be performed at baseline, 24 and 48 weeks. The primary objective will involve calculation of σ and ρ using all data; δ will be estimated by comparing the two alendronate arms pooled to the no-treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 infection
* Adult (aged >18 years or as per local guidelines)
* Premenopausal, if female
* Antiretroviral-naïve
* Starting first-line ART including tenofovir/emtricitabine with either efavirenz (co-formulated as Atripla®) or elvitegravir, cobicistat (co-formulated as Stribild®)
* Low (<10%) ten-year fracture risk as assessed by the FRAX score validated for Canadian populations

Exclusion Criteria:

* Presence of established osteoporosis at baseline as determined by BMD measurement
* Prior or current use of any bone anti-resorptive therapy (eg. bisphosphonate, estrogens with the exception of oral contraceptive pills, etc.)
* Inability to communicate in English
* Creatinine clearance <35 mL/min (using Cockcroft-Gault formula)
* Hypersensitivity to alendronate, other bisphosphonates, or any component of the formulation
* Hypocalcemia
* Abnormalities of the esophagus which delay esophageal emptying such as stricture or achalasia
* Inability to stand or sit upright for at least 30 minutes
* Pregnancy, active plans to become pregnant, or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-04-23 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2018-03-19 (Actual)

PRIMARY OUTCOMES:
Percentage changes in BMD at a) the lumbar spine and b) proximal femur | 48 weeks
  The primary analysis will compare the percentage changes in BMD for the two alendronate/vitamin D arms pooled against the control arm.

SECONDARY OUTCOMES:
Feasibility | 48 weeks
  The proportion of patients who are eligible and who consent to participate will be calculated, and the timeliness (rate) of enrollment will be described, to further inform the feasibility of a larger randomized controlled trial.
Acceptability | 48 weeks
  Using standardized questions, participants will be asked about the acceptability of the alendronate therapy (including the experience of pill-taking and the weekly schedule)
Safety/Tolerability | 48 weeks
  As per Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events.
Adherence | 48 weeks
  Adherence with anti-resorptive therapy will be assessed by pill count and questionnaire.
Bone Biomarkers | 48 weeks
  Two bone biomarkers will be assessed: cross-linked carboxyterminal-telopeptide (CTX) and aminoterminal propeptide of type 1 collagen (P1NP).

CONTACTS AND LOCATIONS:
Overall Officials: Darrell Tan, MD, Principal Investigator — Unity Health Toronto
Locations (2):
- Canada (2):
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario